CLINICAL TRIAL: NCT02737956
Title: The Characteristics and Clinical Outcomes of Acute Myocardial Infarction
Brief Title: The Prognosis of Acute Myocardial Infarction
Acronym: AMI-COPS
Status: Completed | Type: Observational
Sponsor: Xinjiang Medical University (Other)
Responsible Party: Principal Investigator, Xiang Xie, Xiangxie, MD,Professor, The First Affiliated Hospital Of XinJiang Medicial University, Xinjiang Medical University
Other Study IDs: 20160317-03
Record Dates: First submitted 2016-04-05; First posted 2016-04-14 (Estimated); Last update posted 2024-03-28 (Actual); Status verified 2024-03

CONDITIONS: Acute Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- AMI patients with treatment of PCI: All the patiets treat with PCI were enrolled and recorded the clinical characteristic and outcomes during the follow-up period.
- Medication: All the patiets treat with medication (standard secondary prevention) without PCI were enrolled and recorded the clinical characteristic and outcomes during the follow-up period.

SUMMARY:
This study aims to establish a registry and surveillance system for acute myocardial infarction (AMI) patients in Xinjiang, focusing on collecting comprehensive information including basic patient demographics, patient characteristics, diagnostic methods, treatment programs, and hospitalization outcomes such as mortality, treatment complications, hospitalization costs, and follow-up events (death, major adverse cardiac events). The goal is to identify and propose effective prevention strategies to reduce the incidence of AMI, optimize the management and outcomes of AMI patients by implementing guideline recommendations in clinical practice, and conduct analyses to develop effective treatment strategies and predictive models for clinical outcomes. This focus on Xinjiang aims to provide a comprehensive understanding of AMI within this specific geographic and demographic context, ultimately contributing to improved prevention, treatment, and management of AMI patients.

DETAILED DESCRIPTION:
The objective of this study is to establish a comprehensive registry and surveillance system for acute myocardial infarction (AMI) patients in Xinjiang. This platform is designed to support clinical research and translational medicine, aiming to improve the quality of AMI patient care through the integration of guideline recommendations into clinical practice. By collecting detailed information on patient demographics, characteristics, diagnostic methods, treatment programs, and outcomes, including mortality, complications, hospitalization costs, and follow-up events such as death and major adverse cardiac events, this study seeks to lay the foundation for future quality improvement initiatives and research. The ultimate goal is to translate research findings into improved care practices for AMI patients, thereby reducing morbidity and mortality associated with the condition. This endeavor will bridge the gap between clinical research and practical healthcare delivery, ensuring that advancements in the treatment and management of AMI directly benefit patients in Xinjiang, contributing to substantial improvements in healthcare outcomes.

ELIGIBILITY:
Inclusion Criteria:

Acute myocardial infarction patients in hospitalized of the First Affiliated Hospital of Xinjiang Medical University (include diagnosed acute ST-elevation or non ST-elevation myocardial infarction).Diagnosis criteria must meet Universal Definition for AMI (2012).

Exclusion Criteria:

1. Combined with severe valvular heart disease;
2. Combined with severe congenital heart disease;
3. Combined hyperthyroidism, anemia and other high-powered heart disease;
4. With pulmonary heart disease;
5. With hypertrophic obstructive cardiomyopathy;
6. Severe hypotension (SBP <90mmHg or DBP <60mmHg at enrollment);
7. Uncontrolled hypertension (SBP> 160 mmHg before PCI, and / or DBP> 100 mmHg);
8. Liver dysfunction (defined as ALT or total bilirubin is greater than the normal upper limit of 3 times);
9. Renal insufficiency (defined as serum creatinine greater than 1.5 times the normal upper limit);
10. High-risk bleeding patients, such as thrombocytopenia, blood diseases and other diseases;
11. active peptic ulcer and skin ulcers;
12. A patient who is allergic to clopidogrel, tegrellol, or aspirin;
13. Patients with a history of cardiogenic shock within two weeks;
14. pregnant and lactating women, during treatment can not be strict contraception of women of childbearing age;
15. In the past 3 months participated in other clinical researchers;
16. Persons who do not have legal or legal competence;
17. Any condition that the investigator considers unsuitable for participation in the clinical study.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of acute myocardial infarction (AMI) patients hospitalized at the First Affiliated Hospital of Xinjiang Medical University. This includes individuals diagnosed with both acute ST-elevation myocardial infarction (STEMI) and non-ST-elevation myocardial infarction (NSTEMI).
Sampling Method: Probability Sample
Enrollment: 7350 (Actual)
Dates: Start 2012-06-01 (Actual); Primary Completion 2016-05-31 (Actual); Study Completion 2023-12-10 (Actual)

PRIMARY OUTCOMES:
Death | 5 years
  All-cause mortality, Cardiac mortality

SECONDARY OUTCOMES:
Major adverse cardiovascular events (MACE) | 5 years
  Cardiac death, non-fatal myocardial infarction, and target vessel revascularization.
Major adverse cardiovascular and cerebrovascular events (MACCE) | 5 years
  Cardiac death, non-fatal myocardial infarction, target vessel revascularization and stroke.
stroke | 5 years
  ischemic stroke and hemorrhage

CONTACTS AND LOCATIONS:
Overall Officials: Xiang Xie, PhD, Principal Investigator — Xinjiang Medical University
Locations (1):
- First Affilliatted Hospital of Xinjiang Medical University, Ürümqi, Xinjiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yan J, Deng CJ, Wang SF, Aimaitijiang M, Wu TT, Zheng YY, Xie X, Ma YT. Predictive Value of the Modified GRACE Scoring System for All-Cause Mortality in Patients with Acute Myocardial Infarction. Rev Cardiovasc Med. 2023 Jun 6;24(6):161. doi: 10.31083/j.rcm2406161. eCollection 2023 Jun. PMID 39077519
- [Derived] Xiu WJ, Yang HT, Zheng YY, Ma YT, Xie X. Delayed PCI 12 Hours after the Onset of Symptoms Is Associated with Improved Outcomes for Patients with ST-Segment Elevation Myocardial Infarction: A Real-World Study. J Interv Cardiol. 2019 Jun 18;2019:2387929. doi: 10.1155/2019/2387929. eCollection 2019. PMID 31772517